CLINICAL TRIAL: NCT05486689
Title: Evaluation of Physical Activity Before and After Respiratory Rehabilitation in Normal Weight
Brief Title: Evaluation of Physical Activity in Asthmatic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, RicercaTradate, Dr, Istituti Clinici Scientifici Maugeri SpA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2652
Record Dates: First submitted 2022-07-14; First posted 2022-08-03 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Asthma; Physical Activity
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard Program (Experimental): Pulmonary Rehabilitation
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — The enrolled subjects will receivePR program. The 3 weeks inpatient PR will include education, exercise training, nutritional and psychological counselling.
  Education: individualized session of 20 minutes each and group session of 45 minutes each. Endurance training: at least twelve 30-minute daily sessions of supervised incremental exercise training according to Maltais, continuous cycling at 50-70% of the maximal load calculated on the basis of the baseline 6MWT according to Hill. Strength training: twelve 30-minute daily sessions of peripheral limb muscle strength training: 2 set of 8 repetitions during the first week, increased at 12 from the second. The initial load will be set at 30/50% of maximal voluntary isometric strength (MVS). Psychological intervention: individual tailored intervention will be offered when the Hospital Anxiety and Depression Scale (HADS) score is >10 or judged necessary by clinicians, after verifying the subject's motivation.

SUMMARY:
Asthma is a chronic disease, which leads to a number of adverse outcomes, including lower levels of physical activity (PA). Physical inactivity is an important risk factor, increasing PA has become a patient-centred goal for the treatment of subjects with asthma. Data provided by activity monitors are commonly used to measure daily PA.

A recent systematic review showed that adults with asthma had lower levels of total, moderate and vigorous physical activity than those without asthma. There are no data showing the possible effects of a Pulmonary Rehabilitation (PR) program on PA (number of daily steps) in normal-weight subjects with asthma. The main objective of this pilot study is to obtain estimates of the mean value of number of daily steps, time spent on activity in hours and of other variables in normal-weight subjects with asthma measured before and after the PR program. No estimates about these parameters in the same population are currently available from literature search.

DETAILED DESCRIPTION:
Asthma is a chronic disease, which leads to a number of adverse outcomes, including possible lower levels of physical activity (PA). Physical inactivity is an important risk factor, it and was shown that training improves cardiopulmonary fitness, symptoms and quality of life. Increasing PA has become a patient-centred goal for the treatment of subjects with asthma.

Data provided by activity monitors are commonly used to measure daily PA. For PA assessments using an accelerometer, recordings of at least 4 weekly days with a minimum of 8 hours of monitor use (during waking hours) are recommended. A recent systematic review showed that adults with asthma had lower levels of total, moderate and vigorous physical activity than those without asthma. Physical activity appears to be influenced by comorbidities such as obesity in addition to age and sex, decreased disease control, and increased severity. Ather authors involved obese subjects with asthma assigned to a 12-month lifestyle intervention dually targeted modest weight loss (achieve and maintain a weight loss of 7% of baseline body weight) and increased physical activity (achieve and maintain a minimum of 150 minutes per week of moderate intensity physical activity) compared with usual care (control group). Moderately and severely obese adults with uncontrolled asthma showed modest average weight reduction and PA improvements. Finally was showed that a comprehensive pulmonary rehabilitation (PR) program including a weight loss program and exercise training improves PA in moderately-severely obese adults with asthma.

There are no data showing the possible effects of a PR program on PA (number of daily steps) in normal-weight subjects with asthma.

The main objective of this pilot study is to obtain estimates of the mean value (and standard deviation) of number of daily steps, time spent on activity in hours and of other variables in normal-weight subjects with asthma measured before and after the PR program. No estimates about these parameters in the same population are currently available from literature search. This information will be used for formal sample size calculations when planning a future larger study investigating the number of daily steps and time in activity of normal-weight subjects with asthma before and after PR.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of asthma according to GINA step 3-5
* body mass index (BMI) between 18.5 and 24.9 kg/m2
* under optimal medical treatment for at least 3 months according to GINA guideline
* able to perform and complete with studies procedures.

Exclusion Criteria:

* diagnosis of any other chronic pulmonary disease
* smokers or ex-smokers with pack/years ≥10
* acute exacerbation of asthma in the last 30 days
* engagement in exercise training program in the previous 6 months
* history of significant oncological, neurological, cardiovascular diseases
* musculoskeletal impairment
* medical diseases that are likely to compromise mobility and precluding exercise testing and PR
* use of a walker when moving
* reduced spontaneous gait speed (10 m walk test< at 0.8 m/sec).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Physical activity | 5 days after pulmonary rehabilitation
  number of daily steps
Daily activity | 5 days after pulmonary rehabilitation
  hours spent in activity in a day

SECONDARY OUTCOMES:
health-related quality of life | 1 day after pulmonary rehabilitation
  Asthma Quality of Life Questionnaire (AQLQ), 0-7 (higher score indicating better quality of life)
Asthma control | 1 day after pulmonary rehabilitation
  Asthma Control Test (ACT), 5-25 (higher score indicating better asthma control)
Exercise capacity | 1 day after pulmonary rehabilitation
  Six minute walking test (6MWT)
Quadriceps strength | 1 day after pulmonary rehabilitation
  maximal voluntary strength (MVS)
Biceps strength | 1 day after pulmonary rehabilitation
  maximal voluntary strength (MVS)
Mood | 1 day after pulmonary rehabilitation
  Hospital Anxiety and depression scale (HADS), 0-21 0-50 (higher score indicating worst mood)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Visca, Prof, Study Chair — ICS Maugeri
Locations (1):
- Elisabetta Zampogna, Tradate, Va, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliva FM, Tarasconi M, Malovini A, Zappa M, Visca D, Zampogna E. Evaluation of physical activity before and after respiratory rehabilitation in normal weight individuals with asthma: a feasibility study. Front Sports Act Living. 2024 May 9;6:1372048. doi: 10.3389/fspor.2024.1372048. eCollection 2024. PMID 38783863